CLINICAL TRIAL: NCT05886218
Title: A Before/After Study of the Impact of Quantitative Neuromuscular Monitoring and Sugammadex Reversal Following Gastric Bypass Surgery
Brief Title: Quantitative Neuromuscular Monitoring and Gastric Bypass Surgery
Status: Recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 2004503
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-11

CONDITIONS: Sugammadex

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Quantitative Neuromuscular Function Monitoring — Quantitative electromyographic (EMG) monitoring

SUMMARY:
This is a single site, prospective, non-blinded, non-randomized, before/after study. This study is designed to evaluate the impact of monitoring and reversal guidelines for neuromuscular blocking drugs on the post-operative outcomes for patients undergoing laparoscopic gastric bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* scheduled for an elective laparoscopic gastric bypass procedure

Exclusion Criteria:

* age less than 18 years
* pregnancy
* prisoners
* significant co-existing lung disease including asthma or chronic obstructive pulmonary disease (COPD) requiring regular medication
* patients who require supplemental oxygen pre-operatively to maintain a hemoglobin saturation (SpO2>98%)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgical procedures in the UC Davis Medical Center main ORs will be screened for potential enrollment.
Sampling Method: Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Oxygen desaturation | 24 hours
  Incidence and magnitude of significant oxygen desaturation

SECONDARY OUTCOMES:
The rate of compliance with muscle relaxant monitoring and reversal protocols | 24 hours
  Rate of compliance (%)
Total intraoperative rocuronium use | 24 hours
  Total dose/kg/hr (mg/kg/hr)
Total sugammadex dose | 24 hours
  Total dose (mg/kg)
Post-operative supplemental oxygen requirement | 24 hours
  Oxygen requirement (FiO2%/hr)
Post-operative unit length of stay | 7 days
  Length of stay (Hours)
Hospital Length of stay | 7 days
  Length of stay (Hours)
Success rate for wearable device | 24 hours
  Rate of compliance (%)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No